CLINICAL TRIAL: NCT06290414
Title: The Accuracy of Infrared Thermographic Imaging for Assessment of Periodontal Status (A Cross-Sectional Study )
Brief Title: The Accuracy of Infrared Thermographic Imaging for Assessment of Periodontal Status
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shrouk Nabil, Principal Investigator, Ain Shams University
Other Study IDs: FDASU-Rec IM 112318
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases
Keywords: thermography; thermal changes; periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: infrared thermal camera — capturing thermographic imaging of gingiva to detect thermal changes due to inflammation as a result of periodontal disease

SUMMARY:
The diagnosis and differentiation between periodontal diseases are currently based on the measuring and interpretation of full-mouth clinical and radiographic criteria. Thermography is a modern non-invasive imaging method in which the infrared radiation emitted by an object allows the mapping and analysis of the exact temperature distribution on the surface of the object. The produced thermal images correlate with variations in local blood supply and tissue metabolism. Thus, suggested to be a useful rapid and non-invasive tool for the diagnosis of periodontal diseases. However, the validity of this tool compared to standard tools should be evaluated.

DETAILED DESCRIPTION:
A total of 45 of consecutive patients attending the periodontology outpatient clinic will be examined using standard periodontal clinical parameters including; Plaque index (PI), Gingival index (GI), Probing depth (PD), Clinical attachment level (CAL), and standardized periapical radiograph, to identify patients with gingivitis, periodontitis, or healthy periodontium , these 45 patients will be clustered into 3 clusters consisting of 15 patients each to represent each category. The same patients will be examined using an infrared thermal camera (Fluke PTi120 Pocket Thermal Imager), the settings will be all according to the standards of infrared medical diagnosis then the acquired images will be analyzed with (Fluke SmartView IR Analysis Reporting Software and Mobile Application). The images will be interpreted to detect the temperature changes in each mm in tissues in order to determine the patients with gingivitis, periodontitis, or healthy periodontium by an investigator blinded to clinical diagnosis. Then the diagnostic sensitivity and specificity of thermographic images for diagnosis of periodontal diseases will be calculated

ELIGIBILITY:
Inclusion Criteria:

* The patients will be enrolled into the study based on the following inclusion criteria:

  1. Patients with generalized gingivitis
  2. patient with generalized periodontitis .
  3. patient with healthy periodontium .
  4. Both genders above 18 y to 60 y .

Exclusion Criteria:

* The patients will not be enrolled into this study based on the following exclusion criteria:

  1. pregnant women .
  2. smokers .
  3. Patients on medications that cause xerostomia as diuretics , antidepressants

     ,bronchodilators ,antihistaminics , antiepileptic ( etc ..)
  4. Patient using antibiotic, anti-inflammatory, and immunosuppressive therapy during the during the study .
  5. molars according to camera specifications
  6. handicapped patients
  7. para functional habits as mouth breathing and tongue thrusting

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 45 of consecutive patients attending the periodontology outpatient clinic Patients will be selected according to the previously mentioned inclusion and exclusion criteria to be examined clinically and thermographically then they will be clustered into 3 clusters gingivitis , periodontitis and healthy patients based on the clinical diagnosis and each cluster will consist of 15 patients .
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine the agreement of thermographic images for diagnosis of periodontal diseases | 1 day
  Determine the agreement of thermographic images for diagnosis of periodontal diseases through the following outcomes:
  * Sensitivity The proportion of true positives in diseased subjects= True positives/ (true positives + false negatives)
  * Specificity The proportion of true negatives in non-diseased subjects= True negatives/ (true negatives + false positives).

SECONDARY OUTCOMES:
The temperature ranges for healthy periodontium, gingivitis and periodontitis | 1 day
  The temperature ranges for healthy periodontium, and for gingivitis, as well as, for periodontitis will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ola M. Ezzatt, professor, Study Director — faculty of dentistry - Ain Shams University
Locations (1):
- Faculty of dentistry Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Elboray SN, Ezzatt OM, Salah A, Mohamed A, Abdalwahab MM. Evaluation of the Accuracy of Infrared Thermographic Imaging for the Diagnosis of Periodontal Diseases: A Cross-Sectional Study. J Clin Periodontol. 2025 Dec 29. doi: 10.1111/jcpe.70066. Online ahead of print. PMID 41457916